CLINICAL TRIAL: NCT02342483
Title: The Efficacy of the MSM Product on Attenuating Nasal Provocation With a Standardized Allergenic Challenge A Randomized, Double-blind, Adaptive-design Study
Brief Title: MSM Product on Attenuating Nasal Provocation With a Standardized Allergenic Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicus Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: BERG1200
Record Dates: First submitted 2015-01-14; First posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Nasal Breathing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1g (Active Comparator): METHYLSULFONYLMETHANE
  Interventions: Dietary Supplement: MSM
- 3g (Active Comparator): METHYLSULFONYLMETHANE
  Interventions: Dietary Supplement: MSM
- 6g (Active Comparator): METHYLSULFONYLMETHANE
  Interventions: Dietary Supplement: MSM

INTERVENTIONS:
Dietary Supplement: MSM

SUMMARY:
This randomized, double-blind, adaptive design study aims to prove that the Methylsulfonylmethane study product improves nasal breathing and "stuffy nose" symptoms after exposure to environmental allergens. Endpoints include percent change in Peak Nasal Inspiratory Flow, VAS Nasal Symptom Score, number of sneezes and number of used tissues in response to allergen exposure.

DETAILED DESCRIPTION:
Allergic rhinitis, or nasal allergy, is a common condition throughout the world which affects both adult and children alike. It is a group of symptoms characterized by red, itchy eyes, a blocked, itching, runny nose, rhinorrhea, and sneezing. Other reported symptoms include throat clearing, headaches, facial pain, ear pain, itchy throat and palate, snoring, and sleep disturbances. Nasal allergy commonly occurs when an individual's immune system reacts to allergens such as grass, weed, or tree pollens, house dust, mites, mold, and animal dander [1, 2].

Allergic rhinitis is considered to have a substantial effect on the quality of life of a person. Due to the significant effects it demonstrated when left untreated, the disease has gone from being labelled simply as a nuisance to being a serious illness that has to be accounted and medicated. More importantly, such illness was proven to cause asthma and sinusitis [3].

One of the popular nutritional supplements used in treating allergies such as allergic rhinitis, allergic sinusitis, inhalant allergens, and environmental allergens is Methylsulfonylmethane [4].

Methylsulfonylmethane (MSM), also known as dimethyl sulfone and methyl sulfone, is an organic compound containing sulfur that occurs naturally in a variety of fruits, vegetables, grains, and animals, including humans [5]. It is also used in treating arthritis pain, musculoskeletal pain, parasitic infections, rosacea, stretch marks, and alopecia among others [4].

The use of MSM was found to be effective in reducing symptoms of seasonal allergic rhinitis (SAR). It improves the frequency of upper respiratory signs and symptoms such as runny nose, nasal obstruction, and paroxysmal sneezing after a week of oral intake. Furthermore, few side effects were observed, but were not deemed to be of great significance. Thus, MSM was evaluated as a safe medication for SAR [6].

Likewise, MSM administration in rats displayed no adverse events or mortality. No pathological lesions or changes in organ weights were observed [4, 7]. It is proved that MSM is well tolerated in rats and can be a dietary supplement for allergies [4]. In addition, pregnant rats orally administered with MSM showed no adverse effects as well [8]. MSM can be rapidly absorbed, well distributed, and completely disposed from the body 120 hours after initial administration [9].

This randomized, double-blind, adaptive design study aims to prove that the Methylsulfonylmethane study product improves nasal breathing and "stuffy nose" symptoms after exposure to environmental allergens. Endpoints include percent change in Peak Nasal Inspiratory Flow, VAS Nasal Symptom Score, number of sneezes and number of used tissues in response to allergen exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ≥ 18 and ≤ 65 years of age
* Subjects with history of nasal congestion in response to pollen, dust mites, cat dander, and/or dog dander
* Subjects who score "moderate" or "severe" on the VAS Nasal Symptom Score in response to an allergenic challenge at screening (V1)
* Judged by the Investigator to be in general good health on the basis of medical history

Exclusion Criteria:

* Pregnant and/or lactating women
* Subjects with idiopathic rhinitis, atrophic rhinitis, or rhinitis medicamentosa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Peak Nasal Inspiratory Flow (PNIF) | 14 days
VAS Nasal Symptom Score | 14 days
Number of sneezes in response to allergen exposure | 14 days
Number of used tissues in response to allergen exposure | 14 days
Weight of used tissues in response to allergen exposure | 14 days

REFERENCES:
- [Derived] Hewlings S, Kalman DS. Evaluating the Impacts of Methylsulfonylmethane on Allergic Rhinitis After a Standard Allergen Challenge: Randomized Double-Blind Exploratory Study. JMIR Res Protoc. 2018 Nov 29;7(11):e11139. doi: 10.2196/11139. PMID 30497995